CLINICAL TRIAL: NCT06694246
Title: Outpatient Endometrial Biopsy Results; a Quality Improvement Project.
Brief Title: Improving Outpatient Endometrial Biopsy Results
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Al Adan Hospital Kuwait (Industry)
Responsible Party: Principal Investigator, Islam Tarek Elkhateb, Dr, Cairo University
Other Study IDs: QIP2
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Histopathology; Screening Tool; Techniques
Keywords: Pipelle; Endometrial biopsy; histopathology; endometrial sampling; screening; outpatient
MeSH Terms: interventions — Analgesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Endometrial biopsy samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Improving technique — A checklist was developed to ensure the important steps were followed, with tips for obtaining a more adequate sample. This checklist was put in the outpatient procedures room, and each physician performing a biopsy was asked to fill it out.
  Also, a diagram containing illustrative images with the basic steps was put in the procedures room.
  The topic was covered in the biweekly scientific meeting, and all factors attributed to the inadequate sample were discussed.
  The department lead mentioned the topic in the OBGYN department's private messaging group.
  It was finally mentioned in the morning meeting.
Other: Using hysteroscopy in candidate patients — Patients with focal lesions on ultrasound will undergo hysteroscopy and biopsy instead of blind endometrial sampling.
  Patient with stenosed cervix or failed previous sampling might also undergo hysteroscopic guided biopsy.
Other: Analgesia — Analgesia in the form of paracetamol or NSAIDs might be given to some patients 30- 60 minutes before the procedure to reduce the procedure-associated pain and the resultant failure to complete it and obtain an adequate sample.

SUMMARY:
Pipelle is the most commonly used outpatient endometrial biopsy device. Pipelle endometrial biopsy can diagnose 90% of endometrial cancer cases. Pipelle endometrial biopsy is one of the first-line diagnostic procedures for women presenting with abnormal peri- and post-menopausal vaginal bleeding.

Insufficient samples are obtained in 5-23% of cases. In Adan Hospital, a retrospective analysis of all outpatient endometrial samples sent to the histopathology department from April- to October 2024 study showed an insufficient sample percentage of 32% This may be attributed to factors such as patients, equipment, and physicians.

This project aims to improve the endometrial biopsy results by Identifying these factors in the Adan hospital setting, Implementing measures to modify these factors, and finally re-auditing the endometrial biopsy results after six months.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing outpatient endometrial biopsy in the specified time interval (11/2024- 4/2025) will be included.

Exclusion Criteria:

* Could not obtain the sample due to patient physicals, anxiety (patient decline), cervical stenosis, or severe bleeding

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Endometrial biopsy for females with abnormal uterine bleeding
Study Population: All patients undergoing outpatient endometrial sampling
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Adequacy of the sampled endometrial specimen for histopathology diagnosis | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Adan hospital, Kuwait, Al Ahmadi, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided
Patient confidentiality. It may be shared with reasonable request.

REFERENCES:
- [Background] Andrews B, Quick K, MacLeod E, Edwards K, Rone BK. Cervical bleeding with cervical stabilization during IUD placement: allis clamp versus single-tooth tenaculum, a randomized control trial. Arch Gynecol Obstet. 2023 Apr;307(4):1015-1019. doi: 10.1007/s00404-022-06784-x. Epub 2022 Dec 7. PMID 36477274
- [Background] Sierecki AR, Gudipudi DK, Montemarano N, Del Priore G. Comparison of endometrial aspiration biopsy techniques: specimen adequacy. J Reprod Med. 2008 Oct;53(10):760-4. PMID 19004401
- [Background] ACOG Committee Opinion No. 734: The Role of Transvaginal Ultrasonography in Evaluating the Endometrium of Women With Postmenopausal Bleeding. Obstet Gynecol. 2018 May;131(5):e124-e129. doi: 10.1097/AOG.0000000000002631. PMID 29683909
- [Background] ACOG committee opinion no. 557: Management of acute abnormal uterine bleeding in nonpregnant reproductive-aged women. Obstet Gynecol. 2013 Apr;121(4):891-896. doi: 10.1097/01.AOG.0000428646.67925.9a. PMID 23635706
- [Background] Terzic MM, Aimagambetova G, Terzic S, Norton M, Bapayeva G, Garzon S. Current role of Pipelle endometrial sampling in early diagnosis of endometrial cancer. Transl Cancer Res. 2020 Dec;9(12):7716-7724. doi: 10.21037/tcr.2020.04.20. PMID 35117374
- [Background] Blumenthal PD, Berek JS. A Practical Guide to Office Gynecologic Procedures. Lippincott Williams & Wilkins; 2013 Apr 8. Chapter 8
- [Background] Gallos ID, Alazzam M, Clark TJ, Faraj R, Rosenthal AN, Smith PP, Gupta JK. Management of endometrial hyperplasia. Green-top guideline no. 67. RCOG/BSGE Joint Guideline. 2016.
- [Background] Williams PM, Gaddey HL. Endometrial Biopsy: Tips and Pitfalls. Am Fam Physician. 2020 May 1;101(9):551-556. PMID 32352730
- [Background] Del Priore G. Office-based endometrial sampling procedures. In: UpToDate, Connor RF (Ed), Wolters Kluwer. (Accessed on November 28, 2024.)
- Available data/document: Study Protocol — https://drive.google.com/drive/folders/1KXhFMWnU8LAIEVoOEpM2C4iXiE02_8-7?usp=share_link — The above link for inspecting the study protocol and the evidence for a timely study progress.

DOCUMENTS (1):
  • Study Protocol (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT06694246/Prot_000.pdf